CLINICAL TRIAL: NCT05819372
Title: Role of Finite Element Analysis for Selection of Single Point Fixation in Zygomaticomaxillary Complex Fracture
Brief Title: Finite Element and One Point Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, lecturer of oral and maxillofacial surgery, Fayoum University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-OS-2-23-3
Record Dates: First submitted 2023-03-24; First posted 2023-04-19 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Zygomaticomaxillary Complex Fracture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- finite arm (Experimental)
  Interventions: Procedure: Zygomaticomaxillary fracture repair

INTERVENTIONS:
Procedure: Zygomaticomaxillary fracture repair — A cone beam CT (CBCT) scan of the patient will be used to create a 3D scanned image of zygomaticomaxillary complex fracture (ZMC)
  * 3D images will be introduced to finite element (FA) software to evaluate Stresses (MPa), Micromotion (microns), and Life time (cycle) For each model and determine which point of fixation is the best
  * After application this point of fixation on the patient
  * Finite element analysis will be done again to verify the previous results

SUMMARY:
* A cone beam CT (CBCT) scan of the patient, will be used to create a 3D scanned image of ZMC
* 3D images will be introduced to finite element (FA)software to evaluate Stresses (MPa) and Life time (cycle) For each model and determine which point of fixation is the best
* After application this point of fixation on the patient
* Finite element analysis will be done again to verify the previous results

ELIGIBILITY:
Inclusion Criteria:

* Fit to general anesthesia (GA)
* Isolated minimally displaced zygomaticomaxillary complex (ZMC) fracture

Exclusion Criteria:

* absence of other facial trauma, mandibular condylar fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Stresses by megapascal (MPa) | immediately after procedure
  stress on the plate will be measured for each point of application by finite element (FA) software

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, Egypt

REFERENCES:
- [Derived] Refahee SM, Khalifa ME, Askar MG, Breshah MN. Role of finite element analysis for selection of single point fixation in zygomaticomaxillary complex fracture. BMC Oral Health. 2024 Jan 4;24(1):15. doi: 10.1186/s12903-023-03822-1. PMID 38178180